CLINICAL TRIAL: NCT03451942
Title: The Clinical Study of FLOT Regimen Conversion Therapy of Her-2 Negative and Single Site Metastasis Adenocarcinoma of the Stomach / Gastroesophageal
Brief Title: The FLOT Regimen Conversion Therapy of Adenocarcinoma of the Stomach / Gastroesophageal
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, LiuYing, Deputy Chief Physician, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLG-GE-003
Record Dates: First submitted 2018-02-24; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Adenocarcinoma of the Stomach / Gastroesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery group after FLOT regimen chemotherapy (Experimental): After received 4 cycles FLOT regimen chemotherapy , D2 gastric resection and imaging metastases resection was performed. Then continue 4 cycles of FLOT regimen chemotherapy (Chemotherapy begins within 4-6 weeks after surgery)
  Interventions: Drug: FLOT regimen chemotherapy; Procedure: D2 gastric and imaging metastases resection
- FLOT regimen chemotherapy (Placebo Comparator): Continue 4 cycles of the FLOT regimen chemotherapy and evaluate the efficacy every 8 weeks.
  Interventions: Drug: FLOT regimen chemotherapy

INTERVENTIONS:
Drug: FLOT regimen chemotherapy — FLOT regimen chemotherapy
Procedure: D2 gastric and imaging metastases resection — After received 4 cycles FLOT regimen chemotherapy , D2 gastric resection and imaging metastases resection was performed. Then continue 4 cycles of FLOT regimen chemotherapy (Chemotherapy begins within 4-6 weeks after surgery)
  Arms: surgery group after FLOT regimen chemotherapy

SUMMARY:
Evaluate survival benefit of surgical treatment after FLOT regimen conversion therapy of Her-2 Negative and single site metastasis adenocarcinoma of the stomach / gastroesophageal compared with chemotherapy, use relevant biomarkers to evaluate the efficacy of chemotherapy and seek for patients with Her-2 negative and metastatic adenocarcinoma of the stomach / gastroesophageal surviving benefit from surgical treatment after the FLOT regimen conversion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent.
2. Endoscopic biopsy or metastatic biopsy was confirmed to be the adenocarcinoma of the stomach / gastroesophageal.
3. Her - 2 negative(Including: Her protein detection -/1+, and Her protein 2+ but FISH negative).
4. Without any antitumor therapy;
5. According to the 7th edition of AJCC, imaging (CT/MRI) confirmed that the adenocarcinoma of the stomach / gastroesophageal with the initial single site metastasis had a detectable lesion (according to the RECIST 1.1 standard); Single site metastasis includes: liver, spleen, pancreas, ovary, retroperitoneal lymph node (16a1/b2), adrenal gland, kidney;
6. Age from 18 to 70 years.
7. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
8. Life expectancy more than 12 weeks.
9. Histological specimens were provided for biological target detection of her-2;
10. Surgical patients agree to undergo surgery and sign an informed consent to perform the risk of surgery；
11. The main organ function meet the following criteria within 7 days before treatment:

    * blood routine examination( No blood transfusion within 14 days)

      1. HB≥90g/L，
      2. ANC≥1.5×109/L，
      3. PLT≥80×109/L；
    * blood biochemical examination

      1. TBIL <1.5 Upper Limit Of Normal（ULN）;
      2. ALT and AST<2.5ULN(or ≤ 5×ULN in patients with liver metastases).
      3. Cr≤1.5ULN or creatinine clearance>60ml/min.
    * Doppler ultrasonography: left ventricular ejection fraction (LVEF) was lower than normal (50%).
12. Female subjects of child-bearing potential should agree to use contraceptive measures (such as intrauterine contraceptives, contraceptives or condoms) within six months of the study period and the end of the study. The serum or urine pregnancy test was negative within 7 days prior to the study and must be non-lactation. Men subjects should agree to use contraceptives in the study period and within six months at the end of the study period.

Exclusion Criteria:

1. 5 years or at the same time have other malignant tumors；
2. docetaxel or oxaliplatin and other research with chemotherapy drugs are serious allergy;
3. patients with severe cachexia can not eat and can not tolerate chemotherapy and surgery;
4. During the screening period, there was an unknown cause of fever before the first administration and the body temperature was> 38.5 ° C (as judged by the investigators, cancer-related fever subjects could be enrolled);
5. Patients with any severe and / or uncontrollable disease, including:

   1. Patients with hypertension who are not well controlled by antihypertensive medication (systolic BP ≥150 mmHg, diastolic BP ≥100 mmHg);
   2. Myocardial ischemia or myocardial infarction with grade I or above, arrhythmia (including QTc≥480 ms) and ≥2 grade congestive heart failure (New York Heart Association (NYHA) classification);
   3. Severe infection that is active or uncontrollable (≥CTCAE grade 2 infection);
   4. Renal failure requires hemodialysis or peritoneal dialysis;
   5. Have a history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or history of organ transplants;
   6. Poor glycemic control in diabetic patients (fasting blood glucose (FBG)> 10 mmol / L);
   7. Patients with seizures who require treatment;
6. Currently there are gastrointestinal diseases such as intestinal obstruction (including incomplete intestinal obstruction) or the researchers determine the patients may cause gastrointestinal bleeding, perforation or obstruction;
7. Within 4 weeks prior to enrollment, there were non-healing wounds, ulcers or fractures;
8. CNS metastasis;
9. Persons with psychiatric abuse who can not be abdicated or have mental disorders;
10. patients who have participated in other anti-cancer drug clinical trials within 4 weeks;
11. According to the judgment of the researcher, there is a concomitant disease which seriously endangers the safety of the patient or affects the patient in completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Overall survival(OS) | up to 24 months
  the first day of treatment to death or last survival confirm date
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause
R0 resection rate | up to 1 year
  Tumor tissue was completely resected as a percentage of all surgical patients

CONTACTS AND LOCATIONS:
Overall Officials: Ying Liu, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China